CLINICAL TRIAL: NCT04321590
Title: Efficacy of New Products Combining Hydroxycinnamates and Beta-glucans as a Dietary Tool Against Obesity and Associated Dysfunctions (Hyperglycemia and Dyslipemia)
Brief Title: Efficacy of Hydroxycinnamates and Beta-glucans as a Dietary Tool Against obesity_Pilot Study (OBHEALTH_PS)
Acronym: OBHEALTH_PS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Ciencia y Tecnología de Alimentos y Nutrición (Other Government)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Laura Bravo, Professor, Instituto de Ciencia y Tecnología de Alimentos y Nutrición
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AGL2015-69986-R_PS
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Overweight and Obesity
Keywords: Hydroxycinnamates; Beta-glucan; Green coffee bean extract; Dietary supplement
MeSH Terms: conditions — Overweight; Obesity | interventions — beta-glucan, (1-3)(1-4)-

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, double blind study
Who Masked: Participant, Investigator
Masking Description: Blind sachets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3 g 35% beta-glucan (Experimental): Supplement containing 3 g of 35% oat beta-glucan
  Interventions: Dietary Supplement: Combination of oat beta-glucan of different richness (35 and 70%) at low (3g) and high (5g) doses with green coffee bean extract (600 mg)
- 5 g 35% beta-glucan (Experimental): Supplement containing 5 g of 35% oat beta-glucan
  Interventions: Dietary Supplement: Combination of oat beta-glucan of different richness (35 and 70%) at low (3g) and high (5g) doses with green coffee bean extract (600 mg)
- 3 g 70% beta-glucan (Experimental): Supplement containing 3 g of 70% oat beta-glucan
  Interventions: Dietary Supplement: Combination of oat beta-glucan of different richness (35 and 70%) at low (3g) and high (5g) doses with green coffee bean extract (600 mg)
- 5 g 70% beta-glucan (Experimental): Supplement containing 5 g of 70% oat beta-glucan
  Interventions: Dietary Supplement: Combination of oat beta-glucan of different richness (35 and 70%) at low (3g) and high (5g) doses with green coffee bean extract (600 mg)

INTERVENTIONS:
Dietary Supplement: Combination of oat beta-glucan of different richness (35 and 70%) at low (3g) and high (5g) doses with green coffee bean extract (600 mg) — Dose-response study on the effect of two different types of oat beta-glucan with different b-glucan content (35% vs. 70%) in combination with a green coffee bean extract rich in polyphenols. Consumption of 2 sachets/day (providing 3 or 5 g/d beta-glucan plus 600 mg polyphenols) during 6 weeks
  Other Names: 35% oat beta-glucan (PromOat(R)Beta Glucan from Tite&Lile; 70% beta-glucan from Garuda Int. Ltd.; green coffee bean extract from Pharmafoods S-L-

SUMMARY:
Randomized, double blind, parallel study to assess the effect of a dietary supplement combining polyphenols (hydroxycinnamates from green coffee) and a soluble dietary fiber (oat beta-glucans) in obese/overweight subjects.

DETAILED DESCRIPTION:
This pilot study intends to select the best combination of beta-glucan and a green coffee bean phenolic extract. Four different supplements were formulated, containing 3 or 5 g of two types of beta-glucan, with 35% and 70% b-glucan content, together with 600 mg of the green coffee bean extract. Blind sachets were prepared containing half the daily dose of the supplement.

60 overweight/obese male and female volunteers (BMI 25-35 kg/m2, 18-60 y old) were recruited and randomly assigned to one of the four intervention groups. Volunteers were instructed to consume one sachet half an hour before lunch and dinner dissolved in 250 mL water daily during 6 weeks.

At the beginning and at the end of the study, volunteers came to the Human Nutrition Unit at the research center after an overnight fast. Urine and blood samples were obtained, blood pressure was measured and anthropometric measurements were performed. Dietary and physical activity records were collected.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese subjects (BMI 25-35 kg/m2)

Exclusion Criteria:

* Smokers
* Pregnant women
* Medication/consumption of vitamins, dietary supplements, etc.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Anthropometric changes | End of 6-week intervention
  Modification in body weight/percentage body fat

SECONDARY OUTCOMES:
Modification in blood lipids | End of 6-week intervention
  Change in total or LDL-cholesterol levels or triglyceride levels

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bravo, Biologist, Principal Investigator — Research Professor
Locations (1):
- Instituto de Ciencia y Tecnología de Alimentos y Nutrición, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No